CLINICAL TRIAL: NCT04965792
Title: Circulating HPV DNA for Post-treatment Surveillance in HPV-positive Oropharyngeal Squamous Cell Carcinoma
Brief Title: Post-treatment Surveillance in HPV+ Oropharyngeal SCC
Status: Active, not recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Eleni Marie Rettig, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 20-340
Record Dates: First submitted 2021-04-19; First posted 2021-07-16 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: HPV; Oropharyngeal Squamous Cell Carcinoma
Keywords: HPV; Oropharyngeal Squamous Cell Carcinoma; HPV + Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Papillomavirus Infections | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HPV-positive oropharyngeal squamous cell carcinoma (HPV-OPC) Patients: Newly diagnosed HPV-positive oropharyngeal squamous cell carcinoma (HPV-OPC) patients will undergo blood testing for circulating tumor HPV DNA.
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — Blood test

SUMMARY:
In this research study the investigators are examining a blood test to detect HPV DNA in the blood that can possibly detect cancer recurrence earlier than with standard surveillance measures.

DETAILED DESCRIPTION:
This research study involves blood tests to detect HPV DNA at regular time points after treatment for HPV-positive oropharyngeal squamous cell carcinoma (HPV-OPC). Participants may undergo scans based on the results of the blood tests. Study participants will also be asked to complete quality of life questionnaires periodically.

Participation in this study may last for up to 3 years. It is expected that about 150 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed incident or recurrent squamous cell carcinoma of the tonsil or base of tongue (oropharynx) - includes biopsy of any lymph node with clinical evidence of an oropharynx tumor (unknown primary carcinoma in an involved cervical neck lymph node is permitted if high-risk HPV testing is positive on the involved node)
* HPV-associated tumor as defined by one or more : positive p16 immunohistochemistry (>70%) OR in situ hybridization OR PCR-based methods
* Age 18 years or older
* Will undergo oropharyngeal cancer treatment with curative intent
* Ability to understand and the willingness to sign a written informed consent document.
* Baseline positive or detectable ctHPV DNA result in plasma OR detectable corresponding HPV DNA in tumor tissue prior to treatment

Exclusion Criteria:

* Distant metastatic disease (M1, AJCC 8th edition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with HPV-positive oropharynx cancer undergoing curative-intent treatment.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Recurrent disease Rate | Up to 5 years
  The proportion of patients with recurrence first detected by ctHPV DNA will be calculated as a percentage and 95% confidence intervals (CI) established using binomial exact calculation.

SECONDARY OUTCOMES:
Recurrence Detection Predictive Properties | Time from first positive ctHPV DNA test to diagnosis of recurrence, assessed up to 5 years
  Estimate positive and negative predictive value, sensitivity and specificity of ctHPV DNA for subsequent diagnosis of recurrent HPV-OPC
Time to diagnosis of recurrence | Time from first positive ctHPV DNA test to confirmed diagnosis of recurrence, assessed up to 5 years
  The median (IQR) number of months between the first positive ctHPV DNA test to definitive diagnosis of recurrence will be calculated.
Progression-free survival (PFS) | Time from registration to the earlier of progression or death due to any cause, assessed up to 5 years
  Calculated using Kaplan Meier method
Overall survival (OS) | Time from registration to death due to any cause, or censored at date last known alive, assessed up to 5 years
  Calculated using Kaplan Meier method
Quality of Life (QOL) | Pre-study, at 3 and 6 months, then at every other visit for the duration of the study up to 5 years
  QOL will be evaluated using the by Fear of Recurrence Questionnaire-Short Form (score range 6-40; lower score is lower fear of recurrence) and EQ-5D-5L questionnaire (5 questions with score range 1-5 where higher score is worse; and one question with score range 0-100 where higher is better).
Cost Comparison | Up to 5 years
  Projected cost of ctHPV DNA-based compared with standard surveillance

CONTACTS AND LOCATIONS:
Overall Officials: Eleni M Rettig, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Background] Rettig EM, Schoenfeld JD, Miller J, Sargent B, Carey E, Margalit DN, Sehgal K, Sethi RKV, Uppaluri R, Tishler RB, Goguen LA, Annino DJ, Sim ES, Jo VY, Wong KS, Guenette JP, Haddad RI, Hanna GJ. A Prospective Trial of Biomarker-Guided Surveillance for HPV-Positive Oropharynx Cancer Using Plasma Tumor Tissue-Modified Viral HPV DNA. Clin Cancer Res. 2025 May 1;31(9):1605-1614. doi: 10.1158/1078-0432.CCR-24-3053. PMID 39715483